CLINICAL TRIAL: NCT00951704
Title: Evaluating the Quality of Prehospital and In-hospital Cardio-pulmonary Resuscitation - Comparing the Compressions to Concurrent Vital Signs (Invasive Blood Pressure, Cerebral Oxygen Saturation, EtCO2) and Iatrogenic Injuries Associated to Chest Compressions.
Brief Title: Evaluation of the Quality of Cardio-Pulmonary Resuscitation (CPR) in Cardiac Arrest Patients
Status: Completed | Type: Observational
Sponsor: Tampere University Hospital (Other)
Collaborators: Turku University Hospital (Other Government); Uppsala University (Other)
Responsible Party: Sponsor
Other Study IDs: R08116
Record Dates: First submitted 2009-07-31; First posted 2009-08-04 (Estimated); Last update posted 2018-12-13 (Actual); Status verified 2018-12

CONDITIONS: Cardiac Arrest
Keywords: CPR; Tissue Perfusion; invasive arterial pressure; exhaled carbon dioxide; Quality of life; Quality of chest compressions; Epidemiology of sudden cardiac arrest(OHCA)
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Cardiac arrest

SUMMARY:
The prognosis of cardiac arrest patients is generally poor. Recent studies have showed that the high quality of CPR increases the survival after cardiac arrest. Therefore the investigators planned this prospective observational study to determine the epidemiology of sudden cardiac arrest in the prehospital setting of Tampere area, the quality of the CPR, and also the associations between depth and frequency of chest compressions and invasive arterial pressure, EtCO2,cerebral oxygenation and iatrogenic injuries associated to chest compressions 1) in patients resuscitated out of hospital by emergency medical service's (EMS's) personals and 2) in-hospital by hospital resuscitation team members. In addition, the investigators will analyze the effects of the chosen method of resuscitation on critical vital signs (Etco2 and invasive pressures): closed-chest CPR is compared to open-chest CPR, or mechanical CPR with a device (AutoPulse-CPR, Cardio Pump) compared to manual CPR guided with quality CPR device. The results will give the investigators important insights into the haemodynamics of CPR which may guide future strategies for the management of cardiac arrest. The research group is also interested in CPR related injuries and mattress effect. Quality of life after CA is evaluated among survivals and the cause of death among non-survivors.

ELIGIBILITY:
Inclusion Criteria:

* cardiac arrest
* > 18 years of age

Exclusion Criteria:

* < 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult population >18 years of age with cardiac arrest
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2008-11; Primary Completion 2015-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
The success rate of current guidelines (depth and frequency of chest compression, epidemiology) | During the resuscitation
Quality of life after CA | 6 months
  Quality of life after CA is usually fairly good measurement of quality of resuscitation attempt

SECONDARY OUTCOMES:
Invasive arterial pressures, cerebral oxygenation (NIRS), EtCO2 | During the resuscitation
survival of cardiac arrest | hospital discharge

OTHER OUTCOMES:
Change in hemodynamics, Change in cerebral saturation, Change in quality of CPR | During resuscitation

CONTACTS AND LOCATIONS:
Overall Officials: Jyrki Tenhunen, MD, PhD, Study Director — Critical Care Medicine Research Group; Sanna Hoppu, MD, PhD, Principal Investigator — Tampere University Hospital; Marko Sainio, MD, Principal Investigator — Turku University Hospital; Klaus Olkkola, MD, PhD, Study Director — Department of Anesthesiology and Intensive Care, Helsinki University Hospital; Heidi Hellevuo, MD, Principal Investigator — Tampere University Hospital; Piritta Setälä, MD, Principal Investigator — Tampere University Hospital; Ilkka Virkkunen, MD, PhD, Study Director — Tampere University Hospital; Heidi Kangasniemi, MD, Principal Investigator — Tampere University Hospital; Joonas Tamminen, Principal Investigator — Tampere University Hospital
Locations (2):
- Finland (2):
  - Tampere University Hospital, Tampere, Pirkanmaa
  - Department of Anesthesiology and Intensive Care, Turku University Hospital, Turku

REFERENCES:
- [Derived] Kangasniemi H, Setala P, Huhtala H, Kamarainen A, Virkkunen I, Jamsen E, Yli-Hankala A, Hoppu S. Out-of-hospital cardiac arrests in nursing homes and primary care facilities in Pirkanmaa, Finland. Acta Anaesthesiol Scand. 2018 Oct;62(9):1297-1303. doi: 10.1111/aas.13152. Epub 2018 May 29. PMID 29845604
- [Derived] Setala P, Hellevuo H, Huhtala H, Kamarainen A, Tirkkonen J, Hoppu S. Risk factors for cardiopulmonary resuscitation-related injuries sustained during out-of-hospital cardiac arrests. Acta Anaesthesiol Scand. 2018 Oct;62(9):1290-1296. doi: 10.1111/aas.13155. Epub 2018 May 24. PMID 29797706
- [Derived] Setala PA, Virkkunen IT, Kamarainen AJ, Huhtala HSA, Virta JS, Yli-Hankala AM, Hoppu SE. End-tidal carbon dioxide output in manual cardiopulmonary resuscitation versus active compression-decompression device during prehospital quality controlled resuscitation: a case series study. Emerg Med J. 2018 Jul;35(7):428-432. doi: 10.1136/emermed-2017-207103. Epub 2018 May 16. PMID 29769232
- [Derived] Sainio M, Hoppu S, Huhtala H, Eilevstjonn J, Olkkola KT, Tenhunen J. Simultaneous beat-to-beat assessment of arterial blood pressure and quality of cardiopulmonary resuscitation in out-of-hospital and in-hospital settings. Resuscitation. 2015 Nov;96:163-9. doi: 10.1016/j.resuscitation.2015.08.004. Epub 2015 Aug 24. PMID 26310837
- [Derived] Sainio M, Sutton RM, Huhtala H, Eilevstjonn J, Tenhunen J, Olkkola KT, Nadkarni VM, Hoppu S. Association of arterial blood pressure and CPR quality in a child using three different compression techniques, a case report. Scand J Trauma Resusc Emerg Med. 2013 Jul 2;21:51. doi: 10.1186/1757-7241-21-51. PMID 23819769
- [Derived] Sainio M, Kamarainen A, Huhtala H, Aaltonen P, Tenhunen J, Olkkola KT, Hoppu S. Real-time audiovisual feedback system in a physician-staffed helicopter emergency medical service in Finland: the quality results and barriers to implementation. Scand J Trauma Resusc Emerg Med. 2013 Jul 1;21:50. doi: 10.1186/1757-7241-21-50. PMID 23816325
- [Derived] Hoppu S, Sainio M, Huhtala H, Eilevstjonn J, Tenhunen J, Olkkola KT. Blood pressure during resuscitation in man--the effect of pause during rhythm analysis revisited. Resuscitation. 2011 Nov;82(11):1460-3. doi: 10.1016/j.resuscitation.2011.06.005. Epub 2011 Jun 17. PMID 21764499